CLINICAL TRIAL: NCT02762331
Title: Pilot Study to Assess Effect of High Dose Ascorbic Acid (Vitamin C) on Inflammation Reduction in Cardiac Surgery Patients.
Brief Title: High Dose Vitamin C in Cardiac Surgery Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Therapy shown effective by larger studies
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HM20000539
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Disorder of Vitamin C; Atrial Fibrillation; Complications Due to Coronary Artery Bypass Graft; Heart Valve Disease
Keywords: Vitamin C; Coronary Artery Bypass Grafting; Atrial Fibrillation; Cardiac Valve Repair
MeSH Terms: conditions — Atrial Fibrillation; Heart Valve Diseases | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Intravenous ascorbic acid 50 mg/kg in 50 mL normal saline every six hours for 48 hours.
  Interventions: Drug: Ascorbic Acid
- Normal saline (Placebo Comparator): Intravenous normal saline 50 mL every six hours for 48 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ascorbic Acid — Comparing safety and efficacy of IV Vitamin C in CABG patients
  Other Names: Vitamin C
  Arms: Vitamin C
Drug: Placebo — Placebo intervention
  Other Names: Normal Saline
  Arms: Normal saline

SUMMARY:
Coronary artery bypass grafting (CABG) is the most common procedure performed by cardiac surgeons. Post-operative atrial fibrillation (AF) is the most common adverse event following CABG, experienced in 20-50% of patients; the highest incidence of AF occurs by the third post-operative day. Reduction of AF by various drugs is moderately effective, but involves either rate control with beta blockers or rate conversion with amiodarone after the myocardial damage processes initiating AF have already occurred. Decreasing the incidence of post-operative AF, and hence the morbidity and mortality of high-risk CABG patients, could be more fruitfully approached by targeting the upstream combined processes of inflammation and coagulation activation induced by the surgical insult and associated ischemia-reperfusion (I/R). We propose that cell damage induced by oxidative stress and I/R injury could be prevented and/or inhibited by antioxidant supplementation. Specifically the investigators hypothesize that high-dose intravenous (IV) vitamin C supplementation will ameliorate ROS and therefore damp down upstream inflammatory processes, leading to a reduction of downstream adverse events with demonstrable links to inflammation processes, such as AF.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is the most common procedure performed by cardiac surgeons. More complicated surgeries were enabled by the development of cardiopulmonary bypass (CPB) in the 1930s; CABG procedures increased to peak at over 500,000 in 2000, although numbers have decreased somewhat in the last decade. In 2010 over 150,000 major cardiac procedures involved CABG; 18,008 involved both aortic valve replacement and CABG; 2,378 involved mitral valve replacement and CABG; and 4,635 involved mitral valve repair and CABG. This procedure is costly; in 2010 mean hospital charges for CABG and valve procedures were $124,404 and $171,270 with a mean length of hospital stay of 9 and 11 days and an in-hospital death rate of 1.8% and 3.9%, respectively.

Post-operative atrial fibrillation (AF) is the most common adverse event following CABG, experienced in 20-50% of patients; the highest incidence of AF occurs by the third post-operative day. Post-operative AF is associated with overall poorer prognosis resulting 4-fold increase in disabling stroke and cognitive impairment, 3-fold risk of cardiac-related death, and increased length of hospital stay. These risks are increased by the changing composition of the patient population over the last 10 years: patients are older and sicker, and are presenting with more complex disease states and co-morbidities, such as severe coronary artery disease (CAD), congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD), diabetes, previous cardiac surgeries with mechanical support device placements, and complex pharmacological histories. A higher prevalence of AF with increased transfusions among CPB patients has also been reported, suggesting a link with increased plasma load of inflammatory markers and mediators from transfused red cells. Reduction of AF by various drugs is moderately effective, but involves either rate control with beta blockers or rate conversion with amiodarone after the myocardial damage processes initiating AF have already occurred.

Decreasing the incidence of post-operative AF, and hence the morbidity and mortality of high-risk CABG patients, could be more fruitfully approached by targeting the upstream combined processes of inflammation and coagulation activation induced by the surgical insult and associated ischemia-reperfusion (I/R). During CPB, the heart is subjected to ischemic periods of varying duration. The cardiac tissue at that point is electrically resting and its metabolic demands are accordingly low. However, there is also a severely diminished supply of oxygen and nutrients. This results in slow but direct myocardium cellular damage, which increases as ischemia duration increases. However, after reperfusion with oxygenated blood, oxidative stress actually peaks because of accumulated oxidative substrates and cellular depletion of reductive compounds. Cardiac damage related to ischemia-reperfusion will be exacerbated in the presence of co-morbidities, such as diabetes and CAD, which are pathologies with a significant reactive oxygen species (ROS) injury component. High levels of ROS in the myocardium contribute to both electrical and structural remodeling of the cardiac muscle, resulting in the development of AF.

I/R-related oxidative stress and ROS activation contribute to cell damage by modifying protein DNA and phospholipids, resulting in lipid peroxidation and thiol-group oxidation, which in turn are linked to the induction of inflammatory cascades. Lipids are important small-molecule metabolites that have roles in a wide variety of physiological processes. The lipidome of eukaryotic cells contains thousands of lipid entities that structurally and chemically regulate cell membranes, store energy, or are precursors of bioactive metabolites. Defects in lipid regulation and metabolism are therefore significant contributors to disease pathophysiology. In particular, eicosanoids are lipid mediators linking coagulation and inflammatory pathways; intracellular oxidant species are essential mediators in eicosanoids synthesis pathways. Thus lipidomic analyses are a potential novel tool for the identification of drivers of underlying pathogenesis and new diagnostic biomarkers.

During CABG, total peroxide (TP) and oxidative stress index approximately double Increased post-bypass plasma levels of inflammatory markers such as C-reactive protein (CRP) and platelets and leukocyte activation have been observed during CPB. Increases in oxidative stress associated with CPB are correlated with a reduction in total plasma antioxidant capacity. These observations are of interest because an antioxidant is a molecule that inhibits the oxidation of other molecules. Oxidation is a chemical reaction that transfers electrons or hydrogen from a substance to an oxidizing agent. Oxidation reactions can produce free radicals. In turn, these radicals can start chain reactions. When the chain reaction occurs in a cell, it can cause damage or death to the cell. Antioxidants terminate these chain reactions by removing free radical intermediates, and inhibit other oxidation reactions by auto-oxidation; hence antioxidants are often reducing agents. The investigators propose that cell damage induced by oxidative stress and I/R injury could be prevented and/or inhibited by antioxidant supplementation. Specifically the investigators hypothesize that high-dose intravenous (IV) vitamin C supplementation will ameliorate ROS and therefore damp down upstream inflammatory processes, leading to a reduction of downstream adverse events with demonstrable links to inflammation processes, such as AF. Vitamin C is an viable therapeutic candidate because it is a powerful antioxidant with an excellent safety profile, and an emerging history of reducing inflammatory markers in both critically ill and traumatically injured patients. Scattered trials have indicated possible benefits of vitamin C in reducing incidence of post-CABG AF (see Literature search). An antioxidant such as vitamin C acts as a scavenger of intracellular oxidant species; as these are essential mediators in eicosanoids synthesis pathways, it is expected that vitamin C supplementation would decrease the thrombotic potential of eicosanoid-mediated pathways, such as the thromboxane (TBX) production pathway. Impaired cardiac blood flow and clot formation associated with AF contributes to congestive heart failure and stroke; therefore reduction of thrombotic potential is another essential feature for the proposed therapeutic agent.

The proposed pilot study described below represents a marked advance on previously-reported trials in that (a) study design is directed towards minimization of systemic bias, and (b) the investigators will perform simultaneous comparisons of multivariate inflammatory and coagulation profile changes over the immediate post-operative time period when inflammatory changes are expected to be at a maximum. The novelty of this approach is the systems-level analysis of lipids and their interacting moieties; new technology allows for rapid quantitative analysis of over 150 lipid mediators in a sample, time and cost effective manner.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Scheduled for elective non-emergent valve repair or replacement, or multi-vessel CABG surgery
* No known coagulopathy prior to surgery

Exclusion Criteria:

* Emergency cardiac surgery
* Ejection fraction < 35%
* Presence of autoimmune disease or currently receiving immunosuppressant therapy
* History of renal calculi
* Renal dysfunction (pre-operative creatinine clearance < 40 mL/min, or serum creatinine greater than 1.8 mg/dl)
* Known bleeding diathesis
* Active infection, cancer or tumor
* Prior history of atrial fibrillation
* Single CABG procedure (one involved coronary vessel)
* Prisoner
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald F Brophy, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quality AfHRa. HCUPnet: A tool for identifying, tracking, and analyzing national hospital statistics. In: Services DoHaH, ed. Rockville, MD2014.
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):188-97. doi: 10.1161/CIR.0b013e3182456d46. No abstract available. PMID 22215894
- [Background] Surgeons SoT. Adult Cardiac Surgery Database: Executive Summary: 10 Years. 2012; http://www.sts.org/sites/default/files/documents/2012%20-%20AC%20-%203rdHarvestExecutiveSummary.pdf. Accessed January 14, 2014.
- [Background] Korantzopoulos P, Kolettis TM, Galaris D, Goudevenos JA. The role of oxidative stress in the pathogenesis and perpetuation of atrial fibrillation. Int J Cardiol. 2007 Feb 7;115(2):135-43. doi: 10.1016/j.ijcard.2006.04.026. Epub 2006 Jun 9. PMID 16764958
- [Background] Rodrigo R. Prevention of postoperative atrial fibrillation: novel and safe strategy based on the modulation of the antioxidant system. Front Physiol. 2012 Apr 12;3:93. doi: 10.3389/fphys.2012.00093. eCollection 2012. PMID 22518106
- [Background] Mariscalco G, Klersy C, Zanobini M, Banach M, Ferrarese S, Borsani P, Cantore C, Biglioli P, Sala A. Atrial fibrillation after isolated coronary surgery affects late survival. Circulation. 2008 Oct 14;118(16):1612-8. doi: 10.1161/CIRCULATIONAHA.108.777789. Epub 2008 Sep 29. PMID 18824644
- [Background] Fukushima R, Yamazaki E. Vitamin C requirement in surgical patients. Curr Opin Clin Nutr Metab Care. 2010 Nov;13(6):669-76. doi: 10.1097/MCO.0b013e32833e05bc. PMID 20689415
- [Background] Ferguson TB Jr, Coombs LP, Peterson ED; Society of Thoracic Surgeons National Adult Cardiac Surgery Database. Preoperative beta-blocker use and mortality and morbidity following CABG surgery in North America. JAMA. 2002 May 1;287(17):2221-7. doi: 10.1001/jama.287.17.2221. PMID 11980522
- [Background] Halonen J, Hakala T, Auvinen T, Karjalainen J, Turpeinen A, Uusaro A, Halonen P, Hartikainen J, Hippelainen M. Intravenous administration of metoprolol is more effective than oral administration in the prevention of atrial fibrillation after cardiac surgery. Circulation. 2006 Jul 4;114(1 Suppl):I1-4. doi: 10.1161/CIRCULATIONAHA.105.000851. PMID 16820555
- [Background] Wenk MR. The emerging field of lipidomics. Nat Rev Drug Discov. 2005 Jul;4(7):594-610. doi: 10.1038/nrd1776. PMID 16052242
- [Background] Kunt AS, Selek S, Celik H, Demir D, Erel O, Andac MH. Decrease of total antioxidant capacity during coronary artery bypass surgery. Mt Sinai J Med. 2006 Sep;73(5):777-83. PMID 17008938
- [Background] Larmann J, Theilmeier G. Inflammatory response to cardiac surgery: cardiopulmonary bypass versus non-cardiopulmonary bypass surgery. Best Pract Res Clin Anaesthesiol. 2004 Sep;18(3):425-38. doi: 10.1016/j.bpa.2003.12.004. PMID 15212337
- [Background] Review Manager (RevMan) [computer program]. Version Version 5.2. Copenhagen: The Nordic Cochrane Centre; 2012.
- [Background] Higgins JP, Altman DG, Gotzsche PC, Juni P, Moher D, Oxman AD, Savovic J, Schulz KF, Weeks L, Sterne JA; Cochrane Bias Methods Group; Cochrane Statistical Methods Group. The Cochrane Collaboration's tool for assessing risk of bias in randomised trials. BMJ. 2011 Oct 18;343:d5928. doi: 10.1136/bmj.d5928. PMID 22008217

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin C | Normal Saline
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vitamin C: Intravenous ascorbic acid 50 mg/kg in 50 mL normal saline every six hours for 48 hours.
  Ascorbic Acid: Comparing safety and efficacy of IV Vitamin C in CABG patients
  4 subjects total
  Age: Between 32 and 72
  1 Female 3 Male
  1 Black or African American/Non-Hispanic 3 White/Non-Hispanic
  Region of enrollment: USA
- Normal Saline: Intravenous normal saline 50 mL every six hours for 48 hours
  Placebo: Placebo intervention
  2 subjects total
  Age: 50; 74 2 Males 2 White/Non-Hispanic Region of enrollment: USA
- Total: Total of all reporting groups
Arm/Group | Vitamin C | Normal Saline | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Plasma Inflammatory Biomarkers
Description: Change in baseline inflammatory biomarkers including TNF-alpha, C-reactive protein, and interleukin-6 will be measured at 6, 24, and 48 hours following first administration of study drug.
Time Frame: 48 hours
Population: Samples were collected but not analyzed due to study termination. This study was terminated because the therapy was proven effective by larger studies.
Arm/Group | Vitamin C | Normal Saline
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Urinary Inflammatory Biomarker
Description: Change in baseline urine concentrations for neutrophil gelatinase-associated lipocalin (NGAL) will be measured at 6 and 24 hours.
Time Frame: 24 hours
Population: as for outcome 1
Arm/Group | Vitamin C | Normal Saline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Occurence of Atrial Fibrillation
Description: Atrial fibrillation is a common complication of CABG surgery. We will monitor EKG status for development of atrial fibrillation for 48 hours post-op.
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C | Normal Saline
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

4. Secondary Outcome: Coagulation Biomarkers
Description: Change in baseline coagulation biomarkers including thrombomodulin, fibrinogen, platelets and clotting parameters from thromboelastography will be measured at 6, 24, and 48 hours following the first administration of the study drug.
Time Frame: 48 hours
Population: as for outcome 1
Arm/Group | Vitamin C | Normal Saline
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Lipidomic Biomarkers
Description: Change in baseline lipidomic biomarkers including free fatty acids, eicosanoids, 3-polyunsaturated fatty acid-derived lipid mediators, phospholipid substrates of cytosolic PLA2α, and isoprostanes will be measured at 6- and 24 hours following administration of the study drug.
Time Frame: 24 hours
Population: as for outcome 1
Arm/Group | Vitamin C | Normal Saline
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Development of Renal Calculi
Description: We will assess for develop of renal calculi as a safety measure.
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C | Normal Saline
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Investigators will determine daily if any clinical adverse experiences occur during the period from informed consent through study hour 48 and will be followed up through resolution, resolved with sequelae, unresolvable or death.
Description: No adverse events occured
Groups:
- Vitamin C: Intravenous ascorbic acid 50 mg/kg in 50 mL normal saline every six hours for 48 hours.
  Ascorbic Acid: Comparing safety and efficacy of IV Vitamin C in CABG patients
  4 subjects total
  Age: Between 32 and 72
  1 Female 3 Male
  1 Black or African American/Non-Hispanic 3 White/Non-Hispanic
  Region of enrollment: USA No Adverse Events
- Normal Saline: Intravenous normal saline 50 mL every six hours for 48 hours
  Placebo: Placebo intervention
  2 subjects total
  Age: 50; 74 2 Males 2 White/Non-Hispanic
  Region of enrollment: USA No Adverse Events
Arm/Group | Vitamin C | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT02762331/Prot_SAP_000.pdf